CLINICAL TRIAL: NCT01144559
Title: Continuous Femoral Nerve Blocks: Relative Effects of Basal Infusion and Bolus Doses on Sensory and Motor Function
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Brian M. Ilfeld, M.D., M.S./Principal Investigator, University of California, San Diego, Department of Anesthesiology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Femoral Sensory and Motor
Record Dates: First submitted 2010-06-14; First posted 2010-06-15 (Estimated); Last update posted 2010-11-01 (Estimated); Status verified 2010-10

CONDITIONS: Nerve Block
Keywords: Femoral; Nerve Block; Bolus; Continuous Infusion; UCSD; Perineural Catheter; Volunteer; lower extremity nerve blocks

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous Infusion (Active Comparator): Each subject will have one lower extremity (Right or Left) randomized to receive a perineural catheter with a continuous infusion of local anesthetic and then the outcomes will be measured.
  Interventions: Procedure: Continuous Infusion
- Bolus Administration (Active Comparator): The opposite lower extremity (right or left) will be randomized to receive a perineural catheter with the local anesthetic being delivered via a bolus as opposed to continuous as is the case with their other extremity. The outcome measures will then be assessed as described.
  Interventions: Procedure: Bolus Administered

INTERVENTIONS:
Procedure: Continuous Infusion — Extremity randomized continuous infusion will be given a peripheral nerve block and 5cc of Ropivacaine will be administered continuously every hour by a pain pump. Outcome measures will be tested.
  Arms: Continuous Infusion
Procedure: Bolus Administered — Extremity randomized continuous infusion will be given a peripheral nerve block and 5cc of Ropivacaine will be administered using a bolus every hour by a pain pump. Outcome measures will be tested.
  Arms: Bolus Administration

SUMMARY:
This is a research study to determine if the way local anesthetic- or numbing medication- is delivered through a tiny tube next to the nerves that go to the thigh affects the strength and sensation in the thigh.

DETAILED DESCRIPTION:
Specific Aim: Research study to test the null hypothesis that differing the delivery method (continuous basal infusion vs. repeated bolus doses) but providing an equal total dose of Ropivacaine has no impact on quadriceps muscle strength. These results will help define the optimal delivery method of local anesthetic used for continuous peripheral nerve blocks and help guide future research in this clinically relevant area.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* willing to have bilateral femoral perineural catheters place with a subsequent ropivacaine infusion and motor/sensory testing for 9 hours
* willing to stay overnight in the UCSD GCRC/CTRI to allow dissipation of local anesthetic infusion effects by the following morning.

Exclusion Criteria:

* current daily analgesic use
* opioid use with in the previous 4 weeks
* any neuro-muscular deficit of either femoral nerves and/or quadriceps muscles
* pregnancy
* incarceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2010-06; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Quadriceps Femoris Muscle Strength | Every Hour for 14 hours
  The primary end point will be the quadriceps femoris maximum voluntary isometric contraction (MVIC) expressed as percentage of the pre-ropivacaine MVIC: post/pre x 100; with the two sides of each subject compared with each other.
Quadriceps Femoris Muscle Strength | Hour 22
  The primary end point will be the quadriceps femoris maximum voluntary isometric contraction (MVIC) expressed as percentage of the pre-ropivacaine MVIC: post/pre x 100; with the two sides of each subject compared with each other.

SECONDARY OUTCOMES:
Muscle Strength | Every Hour for 14 hours
  This will be evaluated using a portable isometric force dynamometer to measure the maximum voluntary isometric contraction (MVIC) in a seated position.
Sensory Level | Every Hour for 14 hours
  Evaluated in the seated position, using Transcutaneous Electrical Stimulation (TES)in the same manner as outlined in the current anesthesia literature. The current will be increased from 0mA until the subject identifies sensation at which time the current is recorded as the TES value and the nerve stimulator is turned off.
Muscle Strength | Hour 22
  This will be evaluated using a portable isometric force dynamometer to measure the maximum voluntary isometric contraction (MVIC) in a seated position.
Sensory Level | Hour 22
  Evaluated in the seated position, using Transcutaneous Electrical Stimulation (TES)in the same manner as outlined in the current anesthesia literature. The current will be increased from 0mA until the subject identifies sensation at which time the current is recorded as the TES value and the nerve stimulator is turned off.

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Ilfeld, M.D., M.S., Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Medical Center, Hillcrest, San Diego, California, United States